CLINICAL TRIAL: NCT06430255
Title: Effects of Global Postural Re-education Versus Laser-guided Supervised Exercise in Individuals With Non-specific Chronic Low Back Pain: A Randomized Controlled Clinical Trial
Brief Title: Effects of Global Postural Re-education Versus Laser-guided Exercise in Non-specific Chronic Low Back Pain
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Taif University (Other)
Responsible Party: Principal Investigator, Alaa Saleh Baboor, Physical Therapist, Taif University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 24-1243
Record Dates: First submitted 2024-05-16; First posted 2024-05-28 (Actual); Last update posted 2024-05-28 (Actual); Status verified 2024-05

CONDITIONS: Pain, Back
MeSH Terms: conditions — Back Pain

STUDY DESIGN:
Who Masked: Participant
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Global Postural Re-education (Experimental): is a physical therapy method developed in France by Philippe-Emmanuel Souchard. This therapy method is founded on an integrated concept of the muscular system, which is composed of muscle chains. These muscle chains are susceptible to shortening as a result of constitutional, behavioral, and psychological factors, Patients allocated to this group will be having a GPR method course of 8 sessions, two sessions per week for a four-week period. Each session will consist of 3 therapeutic postures, lying, sitting, or standing, to be held for 15-20 minutes each. The postures used are considered the most effective in lengthening the posterior chain, which is usually shortened in patients with LBP.
  Interventions: Other: Global Postural Re-education
- Laser-guided Supervised Exercise (Experimental): Patients allocated to this group will be having a LGSE method course of 8 sessions, two sessions per week for a four-week period. Each session will consist of lumbar movement control exercises. The physiotherapist responsible for the intervention corrected each participant individually as required when performing the movement control exercises to ensure the correct technique. The exercises is progress from the supine position through to standing, 4-point kneeling. The program consists of 8 exercises first starting with abdominal-diaphragmatic breathing and isolated contraction of the transversus abdominis contractions of 10 seconds' duration 5 repetition, Abdominal preparation, Pelvic elevation with previous transversus abdominis contraction and neutral pelvis,
  Interventions: Other: Laser-guided Supervised Exercise

INTERVENTIONS:
Other: Global Postural Re-education — Program for treatment
  Arms: Global Postural Re-education
Other: Laser-guided Supervised Exercise — Program for treatment
  Arms: Laser-guided Supervised Exercise

SUMMARY:
Effects of Global Postural Re-education Versus Laser-guided Supervised Exercise in Individuals With Non-specific Chronic Low Back Pain

DETAILED DESCRIPTION:
The objective of this study will be to investigate the effectiveness of GPR or LGE, in addition to PNE and home exercise program. The primary outcomes will be pain intensity, disability, and fingertip to floor test. The secondary outcomes will be pain catastrophizing, kinesiophobia and depression.

ELIGIBILITY:
Inclusion Criteria:

* Aged between 18 and 45 years.
* Diagnosed with NSLBP.
* Experiencing NSCLBP for ≥ 3 months and score at least 3/10 on the Numerical Pain Rating Scale (NPRS).

Exclusion Criteria:

* Diagnosed with a condition that hinders their ability to engage in physical exercise (e.g., uncontrolled diabetes, cardiovascular disease, orthopedic impairments; balancing problems).
* Diagnosed with severe spine conditions (such as fractures, tumors, ankylosing spondylitis, or inflammatory disorders).
* Diagnosed with neurological problems (such as spine nerve problems or cauda equina syndrome)
* Diagnosed with mental illness or severe cognitive impairment that made it impossible to follow the PNE program.
* With a physical condition that made it impossible to complete the PNE program (the timed "up and go" test had to be completed in 10 seconds at a minimum).
* Receiving alternate therapy for related pathologies (myopathies and neurological diseases) that prevented them from completing the PNE program.

Ages: 18 Years to 45 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 36 (Estimated)
Dates: Start 2024-05-16 (Estimated); Primary Completion 2024-06-25 (Estimated); Study Completion 2024-06-25 (Estimated)

PRIMARY OUTCOMES:
Pain intensity | One month
  assessed using the Numerical Pain Rating Scale which goes from 0 ("no pain at all") to 10 ("worst imaginable pain")
Disability | 7 weeks
  modified Oswestry Low Back Pain Disability (ODI) questionnaire Each part has six statements rated from 0 (least difficult to accomplish action) to 5 (most difficult) The overall score goes from 0 to 50 (the greatest impairment) In individuals with LBP
Fingertip-to-floor test | 7 weeks
  excellent metric properties for LBP

SECONDARY OUTCOMES:
Pain catastrophizing | One month
  will be used to measure pain catastrophizing. Scores range from 0 (never) to 4 (always) for each item (total score = 0-52). Higher ratings reflect more catastrophizing of pain
Kinesiophobia | One month
  will be assessed using the 11 items that make up the TSK-11. The overall score is between 11 and 44 points. A higher score indicates a greater fear of discomfort, movement, and harm.
Depression | 4 weeks
  Patient Health Questionnaire (PHQ-9), The PHQ-9 is a self-administered 9-item questionnaire with four statements ranging from 0 (not at all) to 3 (nearly every day) for each item. A higher total score (20-27) suggests that the patient is suffering from severe depression.

CONTACTS AND LOCATIONS:
Overall Officials: Hosam Alzahrani, Dr, Study Director — Taif University

IPD SHARING:
Plan to Share IPD: No